CLINICAL TRIAL: NCT03616574
Title: Phase 1,Two-part (Dose Escalation, Dose Expansion), Multicenter,Non-randomized,Open-label, Multiple Dose, First-in-human Study of CA102N Monotherapy and of CA102N Combined With Trifluridine/Tipiracil (LONSURF) in Subjects With Advanced Solid Tumors
Brief Title: First-in-human Study of CA102N Monotherapy and CA102N Combined With Trifluridine/Tipiracil (LONSURF) in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Holy Stone Healthcare Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HS-CA102N-101
Record Dates: First submitted 2018-06-26; First posted 2018-08-06 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-03

CONDITIONS: Advanced or Metastatic Solid Tumors; Advanced or Metastatic Colorectal Cancer (mCRC)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Intervention Model Description: Part 1 (dose escalation) of the study will use a conventional 3+3 design (3 subjects per dose cohort, with the potential to add an additional 3 subjects if dose limiting toxicity [DLT] is observed at the same dose level at which the toxicity occurred). Enrollment will occur in 2 groups, CA102N monotherapy (Group A) and CA102N combination therapy (Group B).
  Subjects will be enrolled in Group A first. Once enrollment in Group A has been completed, subsequent subjects will be enrolled in Group B.
  In Part 2 of the study, the safety and tolerability of the preliminary RP2D of CA102N combined with trifluridine/tipiracil (LONSURF) will be further evaluated in up to 12 additional subjects with relapsed or refractory locally advanced or metastatic colorectal cancer who have previously received oxaliplatin and irinotecan-based chemotherapy, an anti-VEGF biological therapy, and if RAS wild-type, an anti-EGFR therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation - CA102N Monotherapy (Experimental): 0.36, 0.54, and 0.72 mg/kg of nimesulide equivalents of CA102N on Days 1 and 15 of a 28-day cycle
  Interventions: Drug: CA102N
- Dose Escalation - CA102N plus LONSURF (Experimental): 0.36, 0.54, and 0.72 mg/kg of nimesulide equivalents of CA102N on Days 1 and 15 in combination with 35 mg/m2/dose of LONSURF orally twice daily on Days 1 through 5 and Days 8 through 12 of each 28-day cycle
  Interventions: Drug: CA102N; Drug: LONSURF
- Dose Expansion - CA102N plus LONSURF (Experimental): The preliminary RP2D of CA102N on Days 1 and 15 in combination with 35 mg/m2/dose of LONSURF orally twice daily on Days 1 through 5 and Days 8 through 12 of each 28-day cycle
  Interventions: Drug: CA102N; Drug: LONSURF

INTERVENTIONS:
Drug: CA102N — CA102N is a covalently bound conjugate of the biological polymer sodium hyaluronate (NaHA) and nimesulide (Nim).
  Other Names: Nim-HA Conjugate
Drug: LONSURF — LONSURF is a cytotoxic combination treatment of 2 new drugs: trifluridine, a thymidine-based nucleoside analog, and tipiracil, an inhibitor of thymidine phosphorylase.
  Other Names: Trifluridine/Tipiracil
  Arms: Dose Escalation - CA102N plus LONSURF; Dose Expansion - CA102N plus LONSURF

SUMMARY:
Study HS-CA102N-101 is a phase 1, two part (dose escalation, dose expansion), multicenter, non-randomized, open-label, multiple dose, first-in-human study of CA102N monotherapy and of CA102N combined with trifluridine/tipiracil (LONSURF) in subjects with advanced solid tumors.

CA102N will be evaluated in subjects with locally advanced or metastatic solid tumours for which no effective therapy is available in Part 1 (dose escalation) and in subjects with relapsed or refractory locally advanced or metastatic colorectal cancer (mCRC) after prior oxaliplatin and irinotecan-based chemotherapy in Part 2 (dose expansion).

DETAILED DESCRIPTION:
Study HS-CA102N-101 is a phase 1, two part (dose escalation, dose expansion), multicenter, non-randomized, open-label, multiple dose, first-in-human study of CA102N monotherapy and of CA102N combined with trifluridine/tipiracil (LONSURF) in subjects with advanced solid tumors.

Part 1 (dose escalation) will determine the safety and tolerability of three dose levels of CA102N as monotherapy and the safety, tolerability and preliminary recommended phase 2 dose (RP2D) of CA102N in combination with trifluridine/tipiracil (LONSURF) in patients with locally advanced or metastatic solid tumors.

Part 2 (dose expansion) will further investigate the safety and tolerability of the combination of CA102N and trifluridine/tipiracil (LONSURF) at the preliminary RP2D in patients with locally advanced or metastatic colorectal cancer that has relapsed after or is refractory to oxaliplatin and irinotecan-based chemotherapy, an anti-vascular endothelial growth factor (VEGF) biological therapy, and if RAS wild-type metastatic colorectal cancer, an anti-epidermal growth factor receptor (EGFR) therapy..

Preliminary efficacy will be evaluated in Parts 1 and 2 of the study as an exploratory endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Subjects enrolled in Part 1 must have histologically documented locally advanced or metastatic solid tumor for which there is no effective therapy available.
* Subjects enrolled in Part 2 must have histologically documented locally advanced or metastatic colorectal cancer that has relapsed after or is refractory to oxaliplatin and irinotecan-based chemotherapy, an anti-VEGF biological therapy, and if RAS wild-type, an anti-EGFR therapy.
* Age ≥18 years (US) or ≥20 years (Taiwan).
* ECOG performance status 0-1.
* Measurable or non-measurable disease based on RECIST version 1.1. Subjects enrolled in Part 2 must have at least one measurable lesion.
* Adequate organ function within 14 days before 1st dose of study drug, defined as:

  1. Platelet count ≥ 100,000/mm3.
  2. Hemoglobin ≥ 9.0 g/dL.
  3. Absolute neutrophil count ≥ 1500/mm3 (without hematopoietic growth factor support).
  4. Creatinine ≤ 1.5 x ULN, or creatinine clearance ≥ 50 mL/min as calculated using the modified Cockcroft-Gault equation.
  5. Aspartate aminotransferase: (i) ≤3 x ULN in subjects without liver metastasis or ≤5 x ULN in subjects with liver metastasis in CA102N monotherapy treatment group; (ii) ≤3 x ULN in subjects who will be treated with CA102N combined with trifluridine/tipiracil (LONSURF).
  6. Alanine aminotransferase: (i) ≤3 x ULN in subjects without liver metastasis or ≤5 x ULN in subjects with liver metastasis in CA102N monotherapy treatment group; (ii) ≤3 x ULN in subjects who will be treated with CA102N combined with trifluridine/tipiracil (LONSURF).
  7. Total bilirubin ≤1.5 x ULN (unless documented Gilbert's Syndrome).
* Has had an adequate treatment washout period prior to 1st dose of study drug defined as:

  1. No major surgery within the past 4 weeks.
  2. No extended field radiation therapy within the prior 4 weeks.
  3. No anticancer therapy or bevacizumab within the prior 3 weeks.
  4. No investigational agent received within prior 4 weeks (or 5 times the half-life of the investigational agent, whichever is shorter).
  5. No aspirin or NSAIDs for at least 72 hours before 1st dose of study drug.
  6. No herbal supplements taken as anticancer agents within the prior 7 days.
* Able to provide written informed consent.
* Life expectancy of ≥ 3 months.
* Women of childbearing potential and men with partners of childbearing potential must agree to use a highly effective means of contraception from study entry through at least 6 months after the last dose of CA102N. Women of childbearing potential are those women who have not been permanently sterilized or are not postmenopausal.

Exclusion Criteria:

* For Part 2, active malignancies other than colorectal cancer.
* History of hypersensitivity or hepatotoxic reaction to nimesulide or to any excipient.
* Requiring therapeutic doses of anticoagulants.
* History or presence of a bleeding tendency or disorder.
* History of gastrointestinal bleed or perforation related to previous NSAID therapy.
* Presence or history of recurrent peptic ulcer or hemorrhage.
* History of cerebrovascular or other active bleeding.
* Myocardial infarction within the last 12 months, severe or unstable angina, symptomatic congestive heart failure New York Heart Association (NYHA) Class III or IV.
* History of a serious cardiac arrhythmia requiring treatment.
* Corrected QT prolongation using Fridericia formula (QTcF), of > 450 msec for males or > 470 msec for females based on a triplicate 12-lead ECG.
* Clinically significant lung disease (eg, interstitial pneumonia, interstitial lung disease, pneumonitis, pulmonary fibrosis, and severe radiation pneumonitis) requiring continuous systemic corticosteroid treatment for 6 months before registration or who are suspected to have such diseases by imaging at Screening.
* Ascites, pleural effusion, or pericardial fluid requiring drainage in last 4 weeks.
* Active autoimmune disease that has required systemic treatment in past 2 years.
* History of allogeneic transplantation requiring immunosuppressive therapy.
* Known positive test for hepatitis B (HBV), hepatitis C (HCV) or human immunodeficiency virus (HIV).
* Clinically active brain metastases, defined as untreated and symptomatic, or requiring therapy with steroids or anticonvulsants to control associated symptoms.
* Pregnant or breast feeding.
* Unresolved toxicity of greater than or equal to NCI-CTCAE (version 5.0) Grade 2 attributed to any prior therapies (excluding anemia, alopecia, skin pigmentation, and platinum-induced neurotoxicity).
* Concomitant medical condition that would increase the risk of toxicity, in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment-related adverse events as assessed by NCI-CTCAE v5.0 | The safety measures will be assessed and recorded throughout the trial until 30 days following treatment termination (an average of 1 year).
  The primary endpoint for the study is the safety and tolerability of CA102N monotherapy and CA102N combined with trifluridine/tipiracil (LONSURF) as determined according to the NCI-CTCAE version 5.0.

SECONDARY OUTCOMES:
Serum concentration of CA102N | Serum sampling timepoints: predose, 0.5,1, 2, 4, 8, 12, 24, 48, and 72 hours postdose CA102N on Days 1 and 15 at Cycle 1 (each cycle is 28 days).
  The secondary endpoint of the study is to measure serum concentration of CA102N (ng/mL).

OTHER OUTCOMES:
Tumor response according to RECIST v1.1 | Tumor response will be evaluated after every 2 cycles of treatment (each cycle is 28 days) until the subject starts alternative anti-cancer treatment or develops progressive disease, whichever occurs first (an average of 1 year).
  The exploratory endpoint of the study is to evaluate objective tumor response to CA102N monotherapy and to CA102N in combination with trifluridine/tipiracil (LONSURF) in subjects with locally advanced or metastatic solid tumors and in subjects with locally advanced or metastatic colorectal cancer. The data of tumor response will be collected and evaluated using RECIST version 1.1.
Analysis of urinary COX-2 metabolites by LC-MS/MS | Urine samples will be collected at predose, 8 and 72 hours postdose CA102N on Days 1 and 15 at Cycle 1, at predose of each subsequent cycle (each cycle is 28 days), until the termination visit (an average of 1 year after Cycle 1 Day 1).
  To determine the systemic alteration of COX-2 metabolites affected by CA102N by analyzing urinary COX-2 metabolites, such as PGEM, PGIM and TXBM, using LC-MS/MS.

CONTACTS AND LOCATIONS:
Overall Officials: Shubham Pant, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jian YS, Chen CW, Lin CA, Yu HP, Lin HY, Liao MY, Wu SH, Lin YF, Lai PS. Hyaluronic acid-nimesulide conjugates as anticancer drugs against CD44-overexpressing HT-29 colorectal cancer in vitro and in vivo. Int J Nanomedicine. 2017 Mar 27;12:2315-2333. doi: 10.2147/IJN.S120847. eCollection 2017. PMID 28392690
- [Derived] Pant S, Dragovich T, Lieu C, Jimeno A, Kundranda M, Menter D, Tchaparian E, Chen YC, Kopetz S. Phase 1 study of the safety, pharmacokinetics, and preliminary efficacy of CA102N as monotherapy and in combination with trifluridine-tipiracil in patients with locally advanced or metastatic solid tumors. Invest New Drugs. 2023 Feb;41(1):25-34. doi: 10.1007/s10637-022-01308-5. Epub 2022 Nov 4. PMID 36331676